CLINICAL TRIAL: NCT03975777
Title: Impact of Exercise Intensity on the Time-course of Mitochondrial Biogenic Gene and Protein Expression in Human Skeletal Muscle.
Brief Title: Time-course of Mitochondrial Biogenic Gene and Protein Expression in Exercised Human Skeletal Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brendon Gurd, PhD (Other)
Responsible Party: Sponsor-Investigator, Brendon Gurd, PhD, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: QMPL-TC-19
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Mitochondrial Biogenesis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-intensity exercise - high-intensity exercise (Experimental): low-intensity exercise session followed by a high-intensity exercise session separated by a minimum of 14 days
  Interventions: Other: LO; Other: HI
- high-intensity exercise - low-intensity exercise (Experimental): high-intensity exercise session followed by a low-intensity exercise session separated by a minimum of 14 days
  Interventions: Other: LO; Other: HI

INTERVENTIONS:
Other: LO — Participants will perform an acute bout of low-intensity cycling (11 x 1 min intervals at ~73% of peak aerobic work rate interspersed with 1 min recovery periods)
Other: HI — Participants will perform an acute bout of high-intensity cycling (8 x 1 min intervals at ~100% of peak aerobic work rate interspersed with 1 min recovery periods)

SUMMARY:
This study examines the impact of exercise intensity on the 12-hour time-course of mitochondrial biogenic gene and protein expression in human skeletal muscle. Briefly, participants will perform two experimental sessions involving an acute bout of work-matched low- or high-intensity interval cycling exercise in a randomized crossover fashion, two weeks apart. Skeletal muscle biopsies will be obtained from the vastus lateralis (3 from each leg) before and 1, 3, 6, 9, and 12 hours post-exercise. Changes in the expression of various transcription factors and mitochondrial proteins will be examined at the mRNA and protein level to determine the time-course of changes in these factors differs between exercise protocols of different intensities.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active (no more than three hours of structured weekly physical activity)
* not currently involved in a systematic training program for improving cardiorespiratory fitness, muscular strength, and/or sport-specific skills
* body mass index < 30 kg/m2

Exclusion Criteria:

* presence of cardiometabolic disease
* taking regular prescription medication for the treatment of cardiometabolic disease
* current cigarette smoker

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in peroxisome proliferator activated receptor (PPAR) gamma co-activator 1-alpha (PGC-1α) messenger ribonucleic acid (mRNA) expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  PGC-1α gene expression (indirect indicator of PGC-1α activity). Transcriptional co-activator involved in the control of mitochondrial biogenesis.

SECONDARY OUTCOMES:
Change in PGC-1α protein content | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  PGC-1α protein content
Change in nuclear factor-erythroid 2 like 2 (Nrf2) mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  Nrf2 gene expression (indirect indicator of Nrf2 activity). Transcription factor involved in the control of mitochondrial biogenesis.
Change in Nrf2 protein content | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  Nrf2 protein content
Change in PPAR-beta mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  PPAR-beta gene expression (indirect indicator of PPAR-beta activity). Transcription factor involved in the control of mitochondrial biogenesis.
Change in estrogen related receptor (ERR)-gamma mRNA expression | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  ERR-gamma gene expression. Transcription factor involved in the control of mitochondrial biogenesis.
Change in leucine-rich pentatricopeptide repeat containing protein 130 (LRP130) mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  LRP130 gene expression. Transcriptional co-activator and RNA-binding protein involved in the transcriptional control and stabilization of mitochondrial mRNAs
Change in LRP130 protein content | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  LRP130 protein content
Change in nuclear respiratory factor-1 (NRF-1) mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  NRF-1 gene expression. Transcription factor involved in the control of mitochondrial biogenesis.
Change in NRF-1 protein content | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  NRF-1 protein content
Change in mitochondrial transcription factor A (TFAM) mRNA expression | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  TFAM gene expression. Transcription factor controlling the expression of mitochondrial-encoded genes.
Change in TFAM protein content | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  TFAM protein content
Change in p53 mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  p53 gene expression. Transcription factor involved in the control of mitochondrial biogenesis.
Change in cytochrome c oxidase subunit 4 (COXIV) mRNA expression. | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  COXIV gene expression. Nuclear encoded subunit of the electron transport chain complex 4 (COX)
Change in COXI mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  COXI gene expression. Mitochondrial encoded subunit of the electron transport chain complex IV (COX)
Change in COXII mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  COXII gene expression.Mitochondrial encoded subunit of the electron transport chain complex IV (COX).
Change in nicotinamide adenine dinucleotide (NADH) subunit 1 (ND1) mRNA expression | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  ND1 gene expression. Mitochondrial encoded subunit of the electron transport chain complex 1 (NADH dehydrogenase)
Change in ND4 mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  ND4 gene expression. Mitochondrial encoded subunit of the electron transport chain complex 1 (NADH dehydrogenase).
Change in citrate synthase (CS) mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  CS gene expression. The first rate limiting enzyme of the Kreb's cycle.
Change in NRF-2 mRNA expression | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  NRF-2 gene expression. Transcription factor involved in the control of mitochondrial biogenesis.
Change in mitochondrial transcription factor B1 (TFB1M) mRNA expression | before exercise to 1, 3, 6, 9, and 12 hours post-exercise
  TFB1M gene expression. Transcription factor controlling the expression of mitochondrial-encoded genes.
Change in mitochondrial transcription factor B2 (TFB2M) mRNA expression | before exercise and 1, 3, 6, 9, and 12 hours post-exercise
  TFB2M gene expression. Transcription factor controlling the expression of mitochondrial-encoded genes.

CONTACTS AND LOCATIONS:
Overall Officials: Brendon J. Gurd, PhD, Principal Investigator — School of Kinesiology and Health Studies
Locations (1):
- School of Kinesiology and Health Studies, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No